CLINICAL TRIAL: NCT06328413
Title: Comparative Evaluation of Pain, Soft Tissue Healing and Density of Newly Formed Bone Tissue in Surgical Extraction Sockets After Leukocyte and Platelet Rich Fibrin and Photobiomodulation Applications
Brief Title: L-PRF vs PBM on Extraction Socket Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Cennet Neslihan Eroglu,DDS,PhD, Assoc Prof Dr, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAEK-302
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Healing Surgical Wounds; Pain
Keywords: photobiomodulation; L-PRF; pain; bone healing; soft tissue healing; third molar
MeSH Terms: conditions — Pain | interventions — Low-Level Light Therapy; Leukocyte Count

STUDY DESIGN:
Intervention Model Description: Since the groups were formed on the same individual, only which side would be the PBM and which side would be the L-PRF group was determined by coin-flip method (simple randomization).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Photobiomodulation group (Experimental): Photobiomodulation application at different extra and intraoral points for 60 seconds with a wavelength of 940 nm in repeated sessions after the extraction of third molar
  Interventions: Device: photobiomodulation
- Leukocyte and platelet-rich fibrin group (Active Comparator): Leukocyte and platelet rich fibrin ( blood product centrifuged for 12 minutes at 2700rpm) application after third molar extraction, single session.
  Interventions: Other: Leukocyte and Platelet Rich Fibrin

INTERVENTIONS:
Device: photobiomodulation — Photobiomodulation application at different extraoral and intraoral points for 60 seconds with a wavelength of 940 nm in repeated sessions after the extraction of third molar
  Arms: Photobiomodulation group
Other: Leukocyte and Platelet Rich Fibrin — Leukocyte and platelet rich fibrin ( blood product centrifuged for 12 minutes at 2700rpm) application after third molar extraction, single session.
  Arms: Leukocyte and platelet-rich fibrin group

SUMMARY:
The aim of this study is to compare leukocyte and platelet-rich fibrin (L-PRF) and photobiomodulation (PBM) applications, which have been repeatedly reported to be superior to control groups, in terms of pain, soft tissue and bone healing in tooth extraction sockets.

DETAILED DESCRIPTION:
After sample size calculation, healthy volunteers were included in the study. Both teeth of these individuals with bilaterally impacted wisdom teeth were extracted simultaneously. Photobiomodulation (PBM) or leukocyte and platelet rich fibrin (L-PRF), an autogenous blood product, was randomly applied to the right or left side extraction sockets. Volunteers were called for repeat sessions (days 2,4,7,7,11,11,14,18 and 21) for the PBM treated side. Follow-ups were performed for pain (days 2,4,7) and soft and bone tissue healing.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class-I healthy volunteers
* Between 18 and 40 years of age who had wisdom teeth (Pell and Gregory Class II, Position B) with bone retention in bilateral symmetrical position with an indication for extraction, and had second molars in the mouth,
* Not use steroids or anti-inflammatory drugs in the last 3 months.

Exclusion Criteria:

* Patients with pericoronitis,
* Smoking habits
* Active periodontal disease
* Pregnancy,
* Breastfeeding
* Unable to give personal consent, and those with missing physical examination and follow-up records were excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Newly formed bone (Healing at extraction sockets) | Bone healing at the end of 1st and 3rd months after third molar extractions
  Newly formed bone assessed on Panoramic x-ray with Image J programme

SECONDARY OUTCOMES:
Soft tissue healing | End of 1st, 2nd week and 1st month after tooth extraction
  Landry Index scores (1: Very poor, 2: Poor, 3: Good, 4. Very Good, 5. Excellent healing)
Probing depth | End of 1st, 2nd week and 1st month after tooth extraction
  Probing depth of second mandibular molar distal pocket (millimeters)

OTHER OUTCOMES:
Postoperative pain | Postoperative 2nd, 4th and 7th days
  Visual Analogue Scale (0=no pain, 10=unbearable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Cennet N Eroglu, DDS,PhD, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No